CLINICAL TRIAL: NCT06841991
Title: The Effect of TeachBack Method on Anxiety and Knowledge Level of Relatives of Patients to Undergo Colonoscopy: A Randomised Controlled Study
Brief Title: Effect of Teach-Back Method in Colonoscopy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Nadiye BARIŞ EREN, Asst. Prof., Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TarsusU-NBARISEREN-002
Record Dates: First submitted 2025-02-14; First posted 2025-02-24 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: Colonoscopy; teach-back; anxiety; education
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teach back education group (Experimental): In the first stage, all participants will be explained about the research and their consent will be obtained. 'Personal Information Form' will be filled out for the relatives of the patients whose informed consents are obtained and who agree to participate in the study. Then, 'Information Questionnaire' and 'State Anxiety Scale' will be administered to all patient relatives as a pretest.
  In the second stage, the relatives of the patients who will undergo colonoscopy will be trained with the Teach-back technique.
  In the third stage, 'Information Questionnaire' and 'State Anxiety Scale' will be applied as posttest after the training. In addition, 'Satisfaction Evaluation of Teach-Back Method' will be performed.
  Interventions: Behavioral: Teach Back Education
- Control Group (No Intervention): In the first stage, all participants will be explained about the research and their consent will be obtained. 'Personal Information Form' will be filled out for the relatives of the patients whose informed consents are obtained and who agree to participate in the study. Then, 'Information Questionnaire' and 'State Anxiety Scale' will be administered to all patient relatives as a pretest.
  No intervention will be made in the second stage. The routine process in the hospital will continue.
  In the third stage, 'Information Questionnaire' and 'State Anxiety Scale' will be administered to the relatives of the patients in both intervention and control groups as posttest after the training.

INTERVENTIONS:
Behavioral: Teach Back Education — The relatives of patients who will undergo colonoscopy will be trained with the teach-back technique.
  Arms: Teach back education group

SUMMARY:
This study aims to evaluate the effect of the training given to the relatives of patients undergoing colonoscopy with the Teach-Back Method on anxiety and knowledge level.

Research hypotheses:

H1: The training given with the Teach-Back Method decreases the anxiety level of patient relatives.

H2: The training provided with the Teach-Back Method increases the knowledge level of patient relatives.

DETAILED DESCRIPTION:
Teach-back technique is an effective educational method that enables a person to rephrase what he/she has learnt in his/her own words to show that he/she understands. There is no study evaluating the effect of the education to be given with the Teach-back technique to the relatives of patients who will undergo colonoscopy. In addition, in this study, anxiety and knowledge levels of the relatives of the patients before and after the training will be discussed and will be a guide for future studies. The training to be given with the Teach-back technique will increase the level of knowledge of the patient's relatives and ensure that they know what to expect at every stage of the procedure. At the end of the study, the participants will be asked about their level of satisfaction with the Teach-back technique. According to the results of the study, it is expected that the use of Teach-back technique in the education of patients and their relatives will increase.

ELIGIBILITY:
Inclusion Criteria:

* To have the ability to communicate verbally,
* Volunteering to participate in the research,
* To be 18 years of age or older.

Exclusion Criteria:

* Lack of verbal communication skills,
* Not volunteering to participate in the research,
* Being under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | 10 minutes
  This form was prepared by the researchers in line with the literature and includes questions questioning the demographic characteristics of the patients' relatives such as age, gender, socioeconomic level, etc. This form will be used before the training
Knowledge Question Form | 20 minutes
  This form consists of questions that will measure the level of knowledge of the patients' relatives about the preparation that should be done before colonoscopy. A literature review will be conducted and 20 multiple-choice questions will be prepared by the researchers. Expert opinion will be obtained from a total of 5 faculty members working in the department of nursing principles in the preparation of this form. Then, the form will be finalised after the necessary arrangements are made. In the form consisting of multiple-choice questions with one correct answer, each question has a value of 5 points. Caregivers can get at least 0 and at most 100 points from the knowledge test. Increasing the score means that the knowledge is sufficient. Questions with incorrect answers are considered as topics to be prioritised in training.
  This form will be used before and after the training.
State Anxiety Inventory | 10 minutes
  This scale was developed by Spielberger and colleagues (1970). The scale was adapted into Turkish by Öner and Le Compte (1998). The scale consists of 20 questions and it is a scale that determines how the individual feels at a certain moment and condition. In the state anxiety scale, the response options collected in four classes are: (1) Not at all, (2) A little, (3) A lot and (4) Completely. The constant value for the State Anxiety Scale is 50. The scores obtained in the state anxiety scale theoretically vary between 20 and 80 points. In the evaluation of the scale, it is accepted that those who score below 36 have no anxiety, those who score between 37 and 42 have mild anxiety and those who score 42 and above have high anxiety.
  This form will be used before and after the training.
Evaluation of Satisfaction with Teach-Back Method | 5 minutes
  The relatives of the patients participating in the study will be asked to give a score between 1-10 in order to determine the level of satisfaction with the training provided by the teach-back method. It is defined as 1-not at all 10- very much and they will be asked to give full points. This form will be used after the training.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oh EG, Lee JY, Lee HJ, Oh S. Effects of discharge education using teach-back methods in patients with heart failure: A randomized controlled trial. Int J Nurs Stud. 2023 Apr;140:104453. doi: 10.1016/j.ijnurstu.2023.104453. Epub 2023 Feb 4. PMID 36827745
- [Background] Oh EG, Lee HJ, Yang YL, Kim YM. Effectiveness of Discharge Education With the Teach-Back Method on 30-Day Readmission: A Systematic Review. J Patient Saf. 2021 Jun 1;17(4):305-310. doi: 10.1097/PTS.0000000000000596. PMID 30882616
- [Background] Eloi H. Implementing teach-back during patient discharge education. Nurs Forum. 2021 Jul;56(3):766-771. doi: 10.1111/nuf.12585. Epub 2021 Apr 30. PMID 33931873
- [Background] Choi S, Choi J. Effects of the teach-back method among cancer patients: a systematic review of the literature. Support Care Cancer. 2021 Dec;29(12):7259-7268. doi: 10.1007/s00520-021-06445-w. Epub 2021 Jul 24. PMID 34302545
- [Background] Ahmadidarrehsima S, Bidmeshki EA, Rahnama M, Babaei K, Afshari M, Khandani BK. The Effect of Self-Management Education by the Teach-Back Method on Uncertainty of Patients with Breast Cancer: a Quasi-Experimental Study. J Cancer Educ. 2020 Apr;35(2):366-372. doi: 10.1007/s13187-019-1474-5. PMID 30680649